CLINICAL TRIAL: NCT02024971
Title: Metact® Combination Tablets Special Drug Use Surveillance Survey on Long-term Use for Type 2 Diabetes Mellitus
Brief Title: Special Drug Use Surveillance of Pioglitazone/Metformin Hydrochloride Combination Tablets Survey on Long-term Use for Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 073-011; JapicCTI-132368 (Registry Identifier: JapicCTI); JapicCTI-R150782 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pioglitazone/Metformin Hydrochloride: Pioglitazone/metformin hydrochloride combination tablets, orally, for 12 months as prescribed by the standard of care.
  Interventions: Drug: Pioglitazone/metformin hydrochloride

INTERVENTIONS:
Drug: Pioglitazone/metformin hydrochloride — Pioglitazone/metformin hydrochloride combination tablets
  Other Names: Metact Combination Tablets

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term use of pioglitazone/metformin hydrochloride combination tablets in the routine clinical setting in patients with type 2 diabetes mellitus for whom therapy with pioglitazone hydrochloride combined with metformin hydrochloride is considered suitable.

DETAILED DESCRIPTION:
This is a special drug use surveillance (survey on long-term use) designed to investigate the safety and efficacy of long-term use of pioglitazone/metformin hydrochloride combination tablets (Metact Combination Tablets) in patients with type 2 diabetes mellitus in the routine clinical setting.

The following items will also be studied:

1. The effects on safety and efficacy caused by changing the administration method of metformin hydrochloride associated with switching to Metact Combination Tablets
2. The effects on compliance associated with switching to Metact Combination Tablets
3. Safety and efficacy in patients who showed inadequate response to pioglitazone hydrochloride and were then switched to Metact Combination Tablets

The planned sample size was 1000 participants. The usual adult dosage is one tablet of Metact administered orally once daily after breakfast (15 mg/500 mg or 30 mg/500 mg of pioglitazone/metformin hydrochloride).

<Precautions Related to Dosage and Administration> Edema due to pioglitazone administration has been reported with comparative frequency in women. Therefore, it is preferable to be vigilant for edema and start Metact Combination Tablets at a dosage equivalent to 15 mg of pioglitazone once daily when administering the study drug to women.

ELIGIBILITY:
Inclusion Criteria:

-Patients with type 2 diabetes mellitus for whom a physician has concluded that therapy with pioglitazone hydrochloride combined with metformin hydrochloride is suitable and for whom long-term treatment with Metact Combination Tablets is considered necessary.

Exclusion Criteria:

-Patients for whom pioglitazone hydrochloride and metformin hydrochloride are contraindicated.

1. Patients with cardiac insufficiency or a history of cardiac insufficiency
2. Patients with the following conditions (i) Patients with a history of lactic acidosis (ii) Dialysis patients (including peritoneal dialysis) (iii) Patients with cardiovascular conditions such as shock, cardiac insufficiency, myocardial infarction, and pulmonary embolism; patients with severely impaired pulmonary function; and patients with other conditions fostering susceptibility to hypoxemia (iv) Patients with excessive alcohol consumption (v) Patients with dehydration (vi) Patients with gastrointestinal disorders such as diarrhea and vomiting (vii) Elderly patients
3. Patients with renal impairment (including mild renal impairment)
4. Patients with hepatic impairment
5. Patients with severe ketosis, diabetic coma or pre-coma, or type I diabetes mellitus
6. Patients with severe infection, severe trauma, or pre- and post-operative patients
7. Patients who are malnourished, starved, debilitated, or have pituitary gland insufficiency or adrenal gland insufficiency
8. Patients with a history of hypersensitivity to the ingredients in Metact Combination Tablets or biguanides
9. Pregnant or potentially pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1103 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 196 investigative sites in Japan from July 2010 to November 2013 (N=1103).
Pre-assignment Details: Patients with type 2 diabetes mellitus for whom a physician has concluded that therapy with pioglitazone hydrochloride combined with metformin hydrochloride is suitable and for whom long-term treatment with Metact Combination Tablets is considered necessary.
Period: Overall Study
Arm/Group | Pioglitazone/Metformin Hydrochloride
Started | 1103
Safety Analysis Set | 1067 (All participants with available data who were enrolled prior to Day 15 of the start of treatment.)
Completed | 1067 (Including 162 patients with missing efficacy data at two or more time points.)
Not Completed | 36
Not completed — Data Not Available | 30
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | Pioglitazone/Metformin Hydrochloride
Number analyzed (Participants) | 1067
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (12.01)
Age, Customized [Number; unit: participants]
  <65 years | 534
  ≥65 years | 533
Age, Customized [Number; unit: participants]
  <20 years | 0
  ≥20 to <30 years | 7
  ≥30 to <40 years | 33
  ≥40 to <50 years | 91
  ≥50 to <60 years | 218
  ≥60 to <70 years | 347
  ≥70 to <80 years | 294
  ≥80 years | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 450
  Male | 617
Pregnancy status (Females) [Number; unit: participants] — Female participants only (n=450)
  participants
    Not pregnant | 450
    Pregnant | 0
Weight [Mean (Standard Deviation); unit: kg] | 69.0 (15.36)
Weight, Customized [Number; unit: participants]
  <40 kg | 7
  ≥40 to <50 kg | 48
  ≥50 to <60 kg | 138
  ≥60 to <70 kg | 193
  ≥70 kg | 310
  Unmeasured | 371
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.61 (4.738)
Body Mass Index, Customized [Number; unit: participants]
  <18.5 kg/m^2 | 10
  ≥18.5 to <25 kg/m^2 | 261
  ≥25 to <30 kg/m^2 | 280
  ≥30 kg/m^2 | 125
  Unknown | 391
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] | 7.5 (6.59)
Duration of Type 2 Diabetes, Customized [Number; unit: participants]
  <2 years | 163
  ≥2 to <5 years | 168
  ≥5 to <10 years | 183
  ≥10 years | 216
  Unknown | 337
Healthcare Category [Number; unit: participants]
  Outpatient | 1049
  Inpatient | 6
  Outpatient and Inpatient | 12
History of Allergies [Number; unit: participants]
  No | 931
  Yes | 95
  Unknown | 41
Presence of Complications [Number; unit: participants]
  No | 132
  Yes | 935
Breakdown of Complications [Number; unit: participants] — Participants may be counted in more than 1 category. DM=diabetes mellitus.
  participants
    Diabetic complications | 169
    Lifestyle-related diseases (excluding DM) | 858
    Liver diseases | 139
    Renal diseases | 9
    Heart or cerebrovascular diseases | 144
    Allergic conditions | 84
    Malignant tumors | 10
    Other | 349
Complications: Breakdown of Diabetic Complications [Number; unit: participants] — Only participants with diabetic complications are reported. Participants may also be counted in more than 1 category.
  participants
    Diabetic nephropathy | 81
    Diabetic retinopathy | 56
    Diabetic neuropathy | 74
Complications: Breakdown of Lifestyle-Related Diseases (Excluding Diabetes Mellitus) [Number; unit: participants] — Participants may be counted in more than 1 category.
  participants
    Hypertension | 656
    Dyslipidaemia | 634
    Hyperuricaemia | 79
Complications: Breakdown of Liver Diseases [Number; unit: participants] — Only participants with liver diseases are reported. Participants may also be counted in more than 1 category.
  participants
    Hepatic steatosis | 107
    Hepatitis alcoholic | 14
    Chronic hepatitis | 17
    Hepatic cirrhosis | 1
Complications: Breakdown of Renal Diseases [Number; unit: participants] — Only participants with renal diseases are reported. Participants may also be counted in more than 1 category.
  participants
    Nephrotic syndrome | 2
    Renal failure chronic | 4
Complications: Breakdown of Heart or Cerebrovascular Diseases [Number; unit: participants] — Only participants with heart or cerebrovascular diseases are reported. Participants may also be counted in more than 1 category.
  participants
    Cardiac failure | 17
    Myocardial infarction | 9
    Angina pectoris | 55
    Cerebral infarction (including late effects) | 52
Stages of Cardiac Failure (New York Heart Association [NYHA] Classification) [Number; unit: participants] — Only participants with cardiac failure are reported. NYHA Class definitions are as follows: Class I - No limitation of physical activity; Class II - Slight limitation of physical activity; Class III - Marked limitation of physical activity; Class IV - Unable to carry on any physical activity without discomfort.
  participants
    Class I | 14
    Class II | 3
    Class III | 0
    Class IV | 0
Complications: Breakdown of Allergic Conditions [Number; unit: participants] — Only participants with allergic conditions are reported. Participants may also be counted in more than 1 category.
  participants
    Asthma bronchial | 33
    Pollinosis | 12
    Rhinitis allergic | 38
    Dermatitis allergic | 11
Complications: Breakdown of Malignant Tumors [Number; unit: participants] — Only participants with malignant tumors are reported. Participants may also be counted in more than 1 category.
  participants
    Gastric cancer | 1
    Large intestine carcinoma | 4
Presence of Medical History [Number; unit: participants] — Breakdown of medical history was categorized as liver disease, renal disease, heart disease, cerebrovascular disease, malignant tumor and any other disease from those mentioned above. Only participants with medical history are presented.
  participants
    No | 875
    Yes | 143
    Unknown | 49
Alcohol History (Drinking Alcohol-Containing Beverages Nearly Every Day) [Number; unit: participants]
  No | 597
  Yes | 293
  Unknown | 177
Smoking Classification [Number; unit: participants]
  Never smoked | 499
  Current smoker | 155
  Ex-smoker | 196
  Unknown | 217
Status of Administration of Pioglitazone and Metformin Prior to Dosing of Metact Combination Tablets [Number; unit: participants]
  Pioglitazone plus metformin prior to dosing | 277
  Pioglitazone alone prior to dosing | 442
  Metformin alone prior to dosing | 211
  Neither pioglitazone nor metformin prior to dosing | 137
Daily Dose of Pioglitazone Prior to Dosing of Metact Combination Tablets [Mean (Standard Deviation); unit: mg/day] | 20.5 (7.60)
Daily Dose of Pioglitazone Prior to Dosing of Metact Combination Tablets [Number; unit: participants] — 348 participants did not take pioglitazone prior to dosing of Metact combination tablet.
  participants
    ≤ 15 mg/day | 456
    > 15 to ≤ 30 mg/day | 258
    > 30 to ≤ 45 mg/day | 5
    > 45 mg/day | 0
Daily Dose of Pioglitazone Before Switching to Metact Combination Tablets,and Metact Dose Assignment [Number; unit: participants] — Metact LD=1 tablet of Metact Combination Tablets low dose. Metact HD=1 tablet Metact Combination Tablets high dose, Pio=Pioglitazone. 348 participants did not take pioglitazone prior to dosing of Metact combination tablet.
  participants
    ≤15 mg/day of Pio to Metact LD | 429
    ≤15 mg/day of Pio to Metact HD | 27
    >15 to ≤30 mg/day of Pio to Metact LD | 46
    >15 to ≤30 mg/day of Pio to Metact HD | 212
    >30 to ≤45 mg/day of Pio to Metact LD | 1
    >30 to ≤45 mg/day of Pio to Metact HD | 4
    >45 mg/day of Pio to Metact LD | 0
    >45 mg/day of Pio to Metact HD | 0
Daily Dose of Metformin Prior to Dosing of Metact Combination Tablets [Mean (Standard Deviation); unit: mg/day] | 681.4 (310.08)
Daily Dose of Metformin Prior to Dosing of Metact Combination Tablets [Number; unit: participants] — Participants may be counted in more than 1 category.
  participants
    < 500 mg/day | 25
    ≥ 500 to < 750 mg/day | 229
    ≥ 750 to < 1500 mg/day | 206
    ≥ 1500 to < 2250 mg/day | 22
    ≥ 2250 mg/day | 6
    ≤ 500 mg/day | 254
    > 500 to ≤ 750 mg/day | 163
    > 750 mg/day | 71
    > 500 mg/day | 234
Daily Dose of Metformin Before Switching to Metact Combination Tablets,and Metact Dose Assignment [Number; unit: participants] — Metact LD=1 tablet of Metact Combination Tablets low dose. Metact HD=1 tablet Metact Combination Tablets high dose, Pio=Pioglitazone. Participants could be counted in more than 1 category. 579 participants did not take Metformin prior to dosing of Metact combination tablet.
  participants
    <500 mg/day of Met to Metact LD | 19
    <500 mg/day of Met to Metact HD | 6
    ≥500 to <750 mg/day of Met to Metact LD | 174
    ≥500 to <750 mg/day of Met to Metact HD | 55
    ≥750 to <1500 mg/day of Met to Metact LD | 155
    ≥750 to <1500 mg/day of Met to Metact HD | 49
    ≥1500 to <2250 mg/day of Met to Metact LD | 12
    ≥1500 to <2250 mg/day of Met to Metact HD | 10
    ≥2250 mg/day of Met to Metact LD | 2
    ≥2250 mg/day of Met to Metact HD | 4
    ≤500 mg/day of Met to Metact LD | 193
    ≤500 mg/day of Met to Metact HD | 61
    >500 to ≤750 mg/day of Met to Metact LD | 124
    >500 to ≤750 mg/day of Met to Metact HD | 37
    >750 mg/day of Met to Metact LD | 45
    >750 mg/day of Met to Metact HD | 26
    Other | 2
Compliance Status of Pioglitazone (Within 3 Months Before Switching to Metact Combination Tablets) [Number; unit: participants] — 348 participants did not take pioglitazone prior to dosing of Metact combination tablet.
  participants
    ≥ 90% | 534
    ≥ 70% | 142
    ≥ 50% | 19
    < 50% | 6
    Unknown | 18
Compliance Status of Metformin (Within 3 Months Before Switching to Metact Combination Tablets) [Number; unit: participants] — 579 participants did not take Metformin prior to dosing of Metact combination tablet.
  participants
    ≥ 90% | 380
    ≥ 70% | 75
    ≥ 50% | 22
    < 50% | 8
    Unknown | 3
Frequency of daily dosing of Metformin prior to dosing of Metact Combination Tablets [Number; unit: participants] — 579 participants did not take Metformin prior to dosing of Metact combination tablet. TID = Three times a day.
  participants
    Daily | 58
    BID | 246
    TID or more | 184
Switch from metformin (> 500 mg/day) to Metact Combination Tablets [Number; unit: participants]
  No | 833
  Yes | 234
Response to pioglitazone in Pioglitazone monotherapy prior to dosing of Metact Combination Tablets [Number; unit: participants] — 625 participants did not take pioglitazone in pioglitazone monotherapy prior to dosing of Metact combination tablet.
  participants
    Inadequate responders | 307 (7.60)
    Patients excluding inadequate responders | 74
    Unknown | 61
Daily dose in Pioglitazone monotherapy prior to dosing of Metact Combination Tablets [Mean (Standard Deviation); unit: mg/day] — Participants who responded poorly to pioglitazone treatment were reported. 760 participants did not take pioglitazone in Pioglitazone monotherapy prior to dosing of Metact combination tablet in patients who responded poorly to pioglitazone treatment.
  mg/day | 20.7 (7.60)
Daily dose in Pioglitazone monotherapy prior to dosing of Metact Combination Tablets [Number; unit: participants] — Participants who responded poorly to pioglitazone treatment were reported. 760 participants did not take pioglitazone in Pioglitazone monotherapy prior to dosing of Metact combination tablet in patients who responded poorly to pioglitazone treatment.
  participants
    ≤ 15 mg/day | 191
    > 15 mg/day to ≤ 30 mg/day | 114
    > 30 mg/day to ≤ 45 mg/day | 2
    > 45 mg/day | 0
Daily dose in Pioglitazone monotherapy prior to switching to Metact Combination Tablets [Number; unit: participants] — Participants who responded poorly to pioglitazone treatment were reported. 760 participants did not take pioglitazone in Pioglitazone monotherapy prior to dosing of Metact combination tablet in patients who responded poorly to pioglitazone treatment.
  participants
    ≤ 15 mg/day of Pio to Metact LD | 178
    ≤ 15 mg/day of Pio to Metact HD | 13
    > 15 mg/day to ≤ 30 mg/day of Pio to Metact LD | 21
    > 15 mg/day to ≤ 30 mg/day of Pio to Metact HD | 93
    > 30 mg/day to ≤ 45 mg/day of Pio to Metact LD | 0
    > 30 mg/day to ≤ 45 mg/day of Pio to Metact HD | 2
    > 45 mg/day of Pio to Metact LD | 0
    > 45 mg/day of Pio to Metact HD | 0
Rate of compliance with the diet regimen at the start of treatment with Metact Combination Tablets [Number; unit: participants]
  ≥ 90% | 270
  ≥ 70% | 367
  ≥ 50% | 259
  < 50% | 76
  Not assessed or compliance status is unknown | 95
Rate of compliance with exercise regimen at the start of treatment with Metact Combination Tablets [Number; unit: participants]
  ≥ 90% | 205
  ≥ 70% | 294
  ≥ 50% | 305
  < 50% | 135
  Not assessed or compliance status is unknown | 128
HbA1c (NGSP value) at the start of treatment with Metact Combination Tablets [Mean (Standard Deviation); unit: percentage of HbA1c] — HbA1c = glycosylated hemoglobin NGSP = National Glycohemoglobin Standardization Program
  percentage of HbA1c | 7.69 (1.369)
Participants with HbA1c (NGSP value) at the start of treatment with Metact Combination Tablets [Number; unit: participants]
  < 6.0% | 39
  ≥ 6.0% to < 7.0% | 270
  ≥ 7.0% to < 8.0% | 340
  ≥ 8.0% | 290
  Unknown | 128
Fasting blood glucose at the start of treatment with Metact Combination Tablets [Mean (Standard Deviation); unit: mg/dL] | 150.1 (56.43)
Participants with Fasting blood glucose at the start of treatment with Metact Combination Tablets [Number; unit: participants]
  < 126 mg/dL | 157
  ≥ 126 to < 140 mg/dL | 75
  ≥ 140 to < 160 mg/dL | 80
  ≥ 160 mg/dL | 134
  Unknown | 621
Fasting insulin at the start of treatment with Metact Combination Tablets [Mean (Standard Deviation); unit: μU/dL] | 10.775 (9.0804)
Participants with Fasting insulin at the start of treatment with Metact Combination Tablets [Number; unit: participants]
  < 1.0 μU/dL | 0
  ≥ 1.0 μU/dL to < 5.0 μU/dL | 24
  ≥ 5.0 μU/dL to < 10.0 μU/dL | 25
  ≥ 10.0 μU/dL to < 50.0 μU/dL | 46
  ≥ 50.0 μU/dL to < 100.0 μU/dL | 1
  ≥ 100 μU/dL | 0
  Unknown | 971

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: 12 months
Population: Safety Analysis Set, all patients for whom data was collected in case report forms, except those who were treated before the contract period, those who were enrolled after Day 15 of the start of treatment with Metact Combination Tablets, and those with missing data after treatment (missed visits).
Measure: Number; unit: participants
Arm/Group | Pioglitazone/Metformin Hydrochloride
Number analyzed (Participants) | 1067
participants
  Thyroid cancer | 1
  Anaemia | 1
  Insomnia | 1
  Dizziness | 2
  Dysgeusia | 1
  Right ventricular failure | 1
  Dyspnoea exertional | 1
  Abdominal distension | 2
  Constipation | 1
  Nausea | 1
  Hepatic function abnormal | 1
  Cold sweat | 1
  Myalgia | 1
  Renal impairment | 1
  Chest discomfort | 1
  Face oedema | 1
  Malaise | 2
  Oedema | 5
  Oedema peripheral | 11
  Cardiothoracic ratio increased | 1
  Blood cholesterol increased | 1
  Blood triglycerides increased | 1
  Lipids abnormal | 1
  Blood creatinine increased | 1
  Weight increased | 4
  Heat illness | 1

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Tabulation of the HbA1c test value and change at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement. n=number of participants analyzed at each time point. Final assessment is defined as a cumulative assessment of Month 12 and Early Termination Visit data.
Time Frame: Baseline and Months 3, 6, 9, 12 and final assessment
Population: The analysis was performed in the efficacy assessment population (n=905).
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Pioglitazone/Metformin Hydrochloride
Number analyzed (Participants) | 905
percentage of HbA1c
  Month 3 (n=819) | -0.47 (1.030)
  Month 6 (n=761) | -0.53 (1.142)
  Month 9 (n=681) | -0.55 (1.183)
  Month 12 (n=670) | -0.60 (1.190)
  Final Assessment (n=896) | -0.58 (1.182)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Tabulation of fasting blood glucose test values and change at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement. n=number of participants analyzed at each time point. Final assessment is defined as a cumulative assessment of Month 12 and Early Termination Visit data.
Time Frame: Baseline and Months 3, 6, 9, 12 and final assessment
Population: The analysis was performed in the efficacy assessment population (n=905).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone/Metformin Hydrochloride
Number analyzed (Participants) | 905
mg/dL
  Month 3 (n=311) | -14.0 (41.98)
  Month 6 (n=275) | -15.5 (40.82)
  Month 9 (n=29) | -11.7 (43.16)
  Month 12 (n=255) | -17.3 (42.97)
  Final Assessment (n=375) | -17.9 (45.36)

4. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: Tabulation of fasting insulin test values and change at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement. n=number of participants analyzed at each time point. Final assessment is defined as a cumulative assessment of Month 12 and Early Termination Visit data.
Time Frame: Baseline and Months 3, 6, 9, 12 and final assessment
Population: The analysis was performed in the efficacy assessment population (n=905).
Measure: Mean (Standard Deviation); unit: μU/dL
Arm/Group | Pioglitazone/Metformin Hydrochloride
Number analyzed (Participants) | 905
μU/dL
  Month 3 (n=22) | -1.768 (4.2928)
  Month 6 (n=46) | -2.374 (7.0954)
  Month 9 (n=22) | -1.018 (5.9072)
  Month 12 (n=51) | -2.524 (9.4260)
  Final Assessment (n=63) | -2.107 (8.7360)

ADVERSE EVENTS:
Time Frame: From baseline to 12 months of treatment.
Description: At each visit the investigator documented occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. The same PTs (Preferred Term) coded for same patient with differing LLTs (Low Level Terms) are counted twice.
Arm/Group | Pioglitazone/Metformin Hydrochloride
Serious Adverse Events (participants affected / at risk) | 18/1067
Other Adverse Events (participants affected / at risk) | 0/1067
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone/Metformin Hydrochloride (N=1067)
Pneumonia (Infections and infestations) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Diabetic hyperglycaemic coma (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Sudden death (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.